CLINICAL TRIAL: NCT07052305
Title: A Phase 1b Study Evaluating the Safety, Tolerability, and Preliminary Anti-tumor Activity of NT-I7 (Efineptakin Alfa), a Long-acting Human IL-7, Post-Axicabtagene Ciloleucel or Post-Lisocabtagene Maraleucel in Subjects With Relapsed/Refractory Large B-cell Lymphoma
Brief Title: NT-I7 (Efineptakin Alfa), a Long-acting Human IL-7, Post-Axicabtagene Ciloleucel or Post-Lisocabtagene Maraleucel in Subjects With Relapsed/Refractory Large B-cell Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: NeoImmuneTech (Industry); The Foundation for Barnes-Jewish Hospital (Other); Daniel E Corbin Lymphoma Research Fund (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202512084
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Large B-cell Lymphoma
Keywords: Non-Hodgkins Lymphoma; Large B-cell Lymphoma; Yescarta; Axi-cel; Breyanzi; Liso-cel; Interleukin 7; NT-I7; CD19 CAR T-cell Therapy
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — efineptakin alfa; Immunotherapy, Adoptive; axicabtagene ciloleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose Escalation Dose Level 1 Starting Dose: NT-I7 (Experimental): NT-I7 will be administered as an intramuscular injection at 600 μg/kg on Day 10 (-2/+5 days) and Day 31 (+/-3 days) post-CAR T-cell therapy infusion, with at least 2 weeks between the NT-I7 injections.
- Dose Escalation Dose Level 2: NT-I7 (Experimental): NT-I7 will be administered as an intramuscular injection at 720 μg/kg on Day 10 (-2/+5 days) and Day 31 (+/-3 days) post-CAR T-cell therapy infusion, with at least 2 weeks between the NT-I7 injections.
- Dose Expansion (RP2D): NT-I7 (Experimental): NT-I7 will be administered as an intramuscular injection at the recommended phase 2 dose on Day 10 (-2/+5 days) and Day 31 (+/-3 days) post-CAR T-cell therapy infusion, with at least 2 weeks between the NT-I7 injections.

INTERVENTIONS:
Drug: NT-I7 — Provided by NeoImmune Tech
  Other Names: Efineptakin alfa
Biological: CAR T-cell therapy — Standard of care: Will be given on day 0 and will be either axicabtagene ciloleucel or lisocabtagene maraleucel .
  Other Names: Axicabtagene ciloleucel; Lisocabtagene maraleucel .

SUMMARY:
Diffuse large B-cell lymphoma is the most commonly occurring subtype of non-Hodgkin lymphoma, but treatment is often not curative, with as many as 50% of patients with adverse risk factors developing relapsed/refractory disease. CAR T-cell therapy has revolutionized modern cancer therapy, with axicabtagene ciloleucel and lisocabtagene maraleucel (anti-CD19 CAR T-cell therapies) FDA approved for second- or later-line treatment of relapsed/refractory large B-cell lymphoma.

IL-7 plays a crucial role in T-cell homeostasis by inducing thymic differentiation, peripheral expansion, and extrathymic differentiation. It is the main regulator of T-cell hemostasis, inducing T-cell growth and proliferation in lymphopenic patients. There is data that suggests that exposure of T-cells to IL-7 may expand T-cells, prevent T-cell exhaustion, and improve effector functions.

NT-I7 is a long-acting human IL-7 cytokine which has been shown in nonclinical studies to increase peripheral T-cells, antitumor efficacy, and tumor infiltrating lymphocytes, either as a monotherapy or in combination with chemo/radiotherapy and/or immune checkpoint inhibitors and CAR T therapy.

This study is testing the hypothesis that the administration of NT-I7 following standard of care (SOC) approved CD19 CAR T-cell therapies for subjects with relapsed/refractory large B-cell lymphoma (LBCL) will be safe and tolerable and may increase the expansion and persistence of CAR T-cells in vivo, which may result in increased tumor response rate and improved clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed relapsed or refractory large B-cell lymphoma, including diffuse large B-cell lymphoma (DLBCL) not otherwise specified (NOS), high grade B-cell lymphoma, DLBCL arising from an indolent lymphoma, grade 3B follicular lymphoma and primary mediastinal large B-cell lymphoma.
* Measurable disease by IWG response criteria for lymphoma.

  * Baseline FDG-PET/CT scan must show FDG-avid lesions compatible with CT-defined anatomical tumor sites.
  * A previously irradiated lesion can be considered a target lesion if it is well defined, measurable, and has clearly progressed following radiation.
  * FDG-PET/CT scans done as SOC up to 60 days pre-lymphodepletion therapy will be allowed. NOTE: After eligibility is confirmed, restaging FDG-PET/CT scans will not be used to change eligibility.
* Eligible for treatment with an FDA-approved SOC CD19 CAR T-cell therapy respective to the current FDA-approved CAR T-cell label for axi-cel(Yescarta®) or liso-cel (Breyanzi®).
* If the patient has previously received an autologous stem cell transplant, s/he must be at least 3 months post-transplant.
* At least 18 years of age.
* ECOG performance status ≤ 2
* Adequate bone marrow and organ function at the start of lymphodepleting chemotherapy as pre-conditioning for SOC CD19 CAR T-cell infusion as defined below:

  * Absolute neutrophil count ≥ 1.0 K/cumm
  * Platelets ≥ 50 K/cumm
  * Hemoglobin ≥ 8.0 g/dL
  * Total bilirubin ≤ 1.5 x IULN or direct bilirubin ≤ IULN for patients with total bilirubin levels > 1.5 x IULN (except for patients with Gilbert's syndrome, who must have a baseline total bilirubin ≤ 3.0 mg/dL)
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x IULN (except for patients with documented liver involvement or bone metastases, who must have an AST and/or ALT ≤ 5.0 x IULN)
  * Alkaline phosphatase ≤ 2.5 x IULN (except for patients with liver metastasis, who must have an alkaline phosphatase ≤ 5.0 x IULN)
  * Creatinine clearance ≥ 30 mL/min by Cockcroft-Gault
  * INR and aPTT ≤ 1.5 x IULN unless the patient is receiving anticoagulant therapy and the PT or aPTT is within the therapeutic range for the anticoagulant. Patients who are on anticoagulation should be able to hold the anticoagulant for 4-5 half-lives of the anticoagulant prior to IM NT-I7 injection to reduce risk of hematoma.
* ECG demonstrating Fridericia's corrected QT interval (QTcF) < 500 ms; patients with QTcF ≥ 500 ms will require clearance by a cardiologist.
* The effects of NT-I7 on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 90 days after the last NT-I7 injection. Should a woman become pregnant or suspect she is pregnant while participating in this study or should a man suspect he has fathered a child, s/he must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.

Exclusion Criteria:

* Previous receipt of an allogeneic solid organ transplant or bone marrow transplant.
* Prior or concurrent malignancy whose natural history has the potential to interfere with the safety or efficacy assessment of the investigational regimen. Patients with prior or concurrent malignancy that does NOT meet that definition are eligible for this trial.
* Chemotherapy or biologic or hormonal therapy for prior or concurrent cancer treatment, within 14 days prior to the first NT-I7 injection.

  * NOTE: Concurrent use of hormones for non-cancer-related conditions (e.g., insulin for diabetes, hormone replacement therapy) is acceptable.
* Currently receiving any other investigational agents, or received within 14 days prior to the first NT-I7 injection.
* Documented active central nervous system (CNS) involvement by lymphoma.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to NT-I7 or other agents used in the study.
* Presence of clinically significant, unresolved toxicities from prior anticancer therapy, defined as having not received to grade ≤ 1 (with the exception of alopecia and laboratory values listed per the inclusion criteria). Patients with irreversible toxicity that is not reasonably expected to be exacerbated by NT-I7 may be included (e.g., hearing loss, peripheral neuropathy) after consultation with the PI.
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection (including active hepatitis A or mycobacterium tuberculosis (testing not required))
  * Congestive heart failure with NYHA Class ≥ 2
  * Uncontrolled atrial fibrillation
  * Any of the following within 6 months prior to day of CAR T-cell administration:

    * Unstable angina pectoris
    * Myocardial infarction
    * Coronary artery bypass grafting
    * Coronary angioplasty
    * Coronary stenting
    * Clinically significant cardiac arrhythmia and/or conduction abnormality
  * Other clinically significant cardiac disease that, in the opinion of the treating physician and/or PI, is a contraindication to study treatment
* History of autoimmune disease for the past 2 years prior to enrollment, including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Bell's palsy, Guillain-Barre syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.

  * NOTE: The following are exceptions to this criterion: vitiligo, alopecia, type 1 diabetes mellitus, autoimmune hypothyroidism stable on hormone replacement, psoriasis not severe enough to require systemic treatment, diverticulitis not associated with inflammatory bowel disease.
* Contraindication to intramuscular therapy.
* Receipt of a live, attenuated vaccine within 30 days prior to NT-I7 injection.

  * NOTE: Patients, if enrolled, should not receive live vaccines during the study period and through 30 days after the last NT-I7 injection. The administration of inactivated vaccines is permitted at any time per the discretion of the treating physician.
* Pregnant and/or breastfeeding and/or expecting to conceive or father children within the study duration (from enrollment through 90 days after last dose of NT-I7). Women of childbearing potential (including women who have had a tubal ligation) must have a negative serum or urine pregnancy test within 72 hours prior to CAR-T administration. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* HIV-infected if not on effective anti-retroviral therapy with undetectable viral load for 6 months. Patients with HIV who are receiving effective anti-retroviral therapy and have had an undetectable viral load for at least 6 months are eligible.
* Evidence of chronic hepatitis B virus (HBV) that is detectable on suppressive therapy. Patients with evidence of chronic HBV infection with undetectable HBV viral load on suppressive therapy are eligible.
* History of hepatitis C virus (HCV) infection that has not been cured or that has a detectable viral load. Patients with a history of HCV that has been treated and cured are eligible. Patients with HCV infection who are currently on treatment and have an undetectable HCV viral load are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-02-10 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | From start of CAR T-cell infusion (day 0) through day 90 (post CAR T-cell infusion)
  Measured per CTCAE v 5.0. CRS and ICANS will be graded per ASTCT guidelines
Maximum tolerated dose of NT-I7 (Dose Escalation only) | From first dose of NT-I7 until 14 days after the second dose NT-I7 dose (estimated to be 35 days)
  Determined by incidence and nature of dose-limiting toxicities (DLTs). DLTs are defined in the protocol.
Recommended phase 2 dose of NT-I7 (Dose Escalation only) | Through 90 days after CAR T-cell infusion
  Determined by the potential correlation of dose levels with safety and efficacy parameters.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Through completion of follow-up (estimated to be 1 year)
  Response will be assessed based on IWG response criteria for lymphoma
Partial response (PR) rate | Through completion of follow-up (estimated to be 1 year)
  Response will be assessed based on IWG response criteria for lymphoma
Complete response (CR) rate | Through completion of follow-up (estimated to be 1 year)
  Response will be assessed based on IWG response criteria for lymphoma
Duration of response (DoR) | Through completion of follow-up (estimated to be 1 year)
  For responders only: defined as the time from the first occurrence of a documented objective response (PR or CR) to the time of the first documented disease progression or death from any cause, whichever occurs first, per IWG.
  Response will be assessed based on IWG response criteria for lymphoma
Progression-free survival (PFS) | Through completion of follow-up (estimated to be 1 year)
  Defined as the time from the CAR T-cell infusion (Day 0) to the first occurrence of progression or death from any cause, whichever occurs first, per IWG.
Overall survival (OS) | Through completion of follow-up (estimated to be 1 year)
  Defined as the time from CAR T-cell infusion (Day 0) to death from any cause.
Effect of NT-I7 on CAR T-cell expansion as measured by quantitative DNA PCR and/or flow cytometry | From day 0 to day 42 post CAR T-cell infusion

CONTACTS AND LOCATIONS:
Overall Officials: Zachary D Crees, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu